CLINICAL TRIAL: NCT03251729
Title: Cervical Cerclage for Preventing Spontaneous Preterm Birth in Singleton Pregnancies Without Prior Spontaneous Preterm Birth and With Short Transvaginal Ultrasound Cervical Length: a Randomized Clinical Trial
Brief Title: Cerclage On LOw Risk Singletons: Cervical Cerclage for Prevention of Spontaneous Preterm Birth in Low Risk Singleton Pregnancies With Short Cervix
Acronym: COLORS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17D.164
Record Dates: First submitted 2017-06-22; First posted 2017-08-16 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Premature Birth
Keywords: cerclage, preterm birth, short cervix
MeSH Terms: conditions — Premature Birth | interventions — Cerclage, Cervical

STUDY DESIGN:
Intervention Model Description: Randomized trial of cerclage versus no cerclage in singleton pregnancies without prior spontaneous preterm birth and with a short transvaginal ultrasound cervical length
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cerclage (Experimental): Cervical cerclage placement along with vaginal progesterone 200mg suppository or 90mg gel nightly from randomization until 36 weeks.
  Interventions: Procedure: Cervical cerclage; Drug: Vaginal progesterone
- Control (Other): Vaginal progesterone 200mg suppository or 90mg gel nightly from randomization until 36 weeks.
  Interventions: Drug: Vaginal progesterone

INTERVENTIONS:
Procedure: Cervical cerclage — Transvaginal cervical cerclage placed between 18 0/7 - 23 6/7 weeks
  Arms: Cerclage
Drug: Vaginal progesterone — Vaginal progesterone 200mg suppository or 90mg gel nightly from randomization until 36 weeks

SUMMARY:
The aim of this study is to evaluate the efficacy of cervical cerclage in prevention of spontaneous preterm birth in singleton pregnancies with a short transvaginal cervical length (<=25mm) and without prior spontaneous preterm birth

DETAILED DESCRIPTION:
Singleton pregnancies between 18 0/7 to 23 6/7 weeks without a prior spontaneous preterm birth found to have a short transvaginal ultrasound cervical length (<=25mm) and meeting all other eligibility criteria will be randomized to either cervical cerclage or control (no cerclage). Aside from cerclage placement, management of included women will be the same including recommendation for daily vaginal progesterone 200mg suppository or 90mg gel from randomization until 36 6/7 weeks. The primary outcome will be the incidence of spontaneous preterm birth <35 weeks

ELIGIBILITY:
Inclusion Criteria:

* 18 year old or older
* Singleton pregnancy
* No prior SPTB or second trimester losses between 160 and 366 weeks
* TVU CL ≤25mm between 180 and 236 weeks

Exclusion Criteria:

* Multiple pregnancy
* Prior SPTB or second trimester losses between 160 and 366 weeks
* Cerclage in situ
* Painful regular uterine contraction and/or preterm labor
* Rupture membranes
* Major fetal anomaly or aneuploidy
* Active vaginal bleeding
* Placenta previa and/or accreta
* Cervical dilation >1.0 cm and/or visible membranes by pelvic exam
* Suspicion of chorioamnionitis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients must be pregnant to be enrolled. Self-represented gender identity is NOT a basis of eligibility
Enrollment: 93 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Preterm birth <35 weeks | At delivery
  Incidence of spontaneous preterm birth less than 35 weeks

SECONDARY OUTCOMES:
Preterm birth <37 weeks, <34 weeks, <32 weeks, <28 weeks, <24 weeks | At delivery
Mean gestational age at delivery | At delivery
Histologically proven clinical chorioamnionitis | At delivery
Neonatal outcomes: birth weight | At delivery
Neonatal outcomes: low birth weight (<2500g), | At delivery
Neonatal outcomes: admission to intensive care nursery | At delivery
Neonatal outcomes: length of neonatal hospital admission | at least 30 days after delivery, up to 6 months after delivery
Neonatal outcomes: respiratory distress syndrome | at least 30 days after delivery, up to 6 months after delivery
Neonatal outcomes: IVH grade 3 or 4 | at least 30 days after delivery, up to 6 months after delivery
Neonatal outcomes: retinopathy of prematurity | at least 30 days after delivery, up to 6 months after delivery
Neonatal outcomes: bronchopulmonary dysplasia | at least 30 days after delivery, up to 6 months after delivery
Neonatal outcomes: neonatal mortality | 28 days after delivery

CONTACTS AND LOCATIONS:
Locations (3):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States
- Italy (2):
  - University of Naples Federico II, Naples
  - University Cattolica del S. Cuore, Rome

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon completion of appropriate data sharing agreements
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1yr after study completion
Access Criteria: IPD will be shared upon completion of appropriate data sharing agreements

REFERENCES:
- [Background] Berghella V, Ciardulli A, Rust OA, To M, Otsuki K, Althuisius S, Nicolaides KH, Roman A, Saccone G. Cerclage for sonographic short cervix in singleton gestations without prior spontaneous preterm birth: systematic review and meta-analysis of randomized controlled trials using individual patient-level data. Ultrasound Obstet Gynecol. 2017 Nov;50(5):569-577. doi: 10.1002/uog.17457. Epub 2017 Oct 5. PMID 28295722
- [Derived] Boelig RC, Tersigni C, Di Simone N, Saccone G, Facchinetti F, Scambia G, Berghella V. Cerclage in singleton pregnancies with no prior spontaneous preterm birth and short cervix: a randomized controlled trial. Am J Obstet Gynecol MFM. 2025 Apr;7(4):101602. doi: 10.1016/j.ajogmf.2025.101602. Epub 2025 Jan 27. PMID 39880123